CLINICAL TRIAL: NCT03154736
Title: Scaling-up Packages of Interventions for Cardiovascular Disease Prevention in Selected Sites in Europe and Sub-Saharan Africa: An Implementation Research
Acronym: SPICES_PHASE_1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Collaborators: ERCR SPURBO (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 29BRC17.0015 SPICES_PHASE_1
Record Dates: First submitted 2017-05-11; First posted 2017-05-16 (Actual); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Cardiovascular Disease
Keywords: CVD; FDRCV; Developing countries; Rcih countries
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Interviews as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interview (Experimental): Individual interview an in a group interview. Socio-economic questionnaire
  Interventions: Other: Interview

INTERVENTIONS:
Other: Interview — Individual interview and group interview Socio-economic questionnaire

SUMMARY:
Cardiovascular disease is the leading cause of death in the world. 17.5 million people died in 2012 due to a cerebrovascular disease (31% of all causes of death). In Europe more than 50% of deaths are due to cardiovascular disease. The mortality rate for cardiovascular disease is higher in the lower socio-economic levels. Three-quarters of deaths from cardiovascular disease occur in developing countries. According to estimates in 2030, cardiovascular disease will be responsible for more deaths than the sum of infectious, nutritional, maternal and perinatal diseases in developing countries.

Measures to prevent cardiovascular risk factors have been shown to be effective.

The lack of an adequate primary care network in developing countries limits the screening and treatment of patients with cardiovascular risk factors. As a result, these patients do not benefit from adequate prevention, are diagnosed late and remain disabled or die at a young age, resulting in significant additional costs for families but also at the macroeconomic level.

Interventions are possible on a large scale (policies against tobacco and adverse dietary behavior, promote physical activity, etc.). Actions are possible on an individual level, both in primary prevention (control of cardiovascular risk factors) and secondary prevention, where many treatments have proved their effectiveness. These interventions are effective and cost-effective from a macroeconomic perspective. It was estimated that the cost of such interventions would not exceed 4% of health expenditure in developing countries and 1-2% in rich countries.

The World Health Organization insists on the importance of the triad composed by the patient and his family, community and health professionals. Results are possible only when these three components work together for the same purpose. Numerous studies show the benefit of the involvement of patients in their care in the rich countries and in the developing countries.

DETAILED DESCRIPTION:
This project builds on advances in the treatment of HIV / AIDS in Sub-Saharan Africa and in chronic disease management through the WHO Innovative Care for Chronic Conditions Framework.

These projects emerged from the observation that the rich country model of care (patient-centered, hospital-centered and specialist approach with regular clinical and paraclinic follow-up) was not transferable to developing countries, The limitation of human, technical and financial resources.

A paradigm shift is needed to improve cardiovascular disease control in a more cost-effective manner.

The SPICES project plans to integrate the current knowledge of new studies to improve the prevention and control of cardiovascular disease in high-, middle-, and low-income countries.

Rich countries and developing countries will therefore be involved in the study: the selected sites are France, the United Kingdom, Belgium, South Africa and Uganda.

This study is a stage of observation in the different countries which will make it possible to make an inventory of the places and to target the most adapted interventions.

The main objective is to define the representations on cardiovascular prevention and the follow up of patients with cardiovascular disease or FDRCV.

The secondary objectives are to identify:

* the brakes in the management of patients with CVD or FDRCV
* the institutional care network for these patients
* Identify the "informal" care network, that is, family and community caregivers and within them the potential barriers and facilitators to their care.

ELIGIBILITY:
Inclusion Criteria:

* Persons aged over 18 years.
* Persons able to express their consent
* Patients with FDRCV or CVD who gave written consent to participate in the study.
* Family caregiver of patients with FDRCV or CVD with written consent to participate in the study

Exclusion Criteria:

* Refusal to participate in the study
* Patients and / or family caregiver who can not express their consent (illiterate, severe cognitive or psychiatric disorders)
* Patients under judicial protection (guardianship and curatorship)
* Pregnant women
* Patients under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2017-10-02 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Experiences of patients with cardiovascular disease | 1 day
  The representations on cardiovascular prevention and the follow-up experience of patients with cardiovascular disease or CVRF will be defined by questionnaire

SECONDARY OUTCOMES:
The obstacles of patients with cardiovascular disease | 1 day
  The obstacles to the management of patients with CVD or CVRF will be identified by questionnaire
Institutional care network | 1 day
  The institutional care network for these patients will be identified by questionnaire
Informal or informal care network | 1 day
  The "informal" care network, that is to say, family or community caregivers and within them the brakes and facilitators will be identified by questionnaire

CONTACTS AND LOCATIONS:
Locations (21):
- France (21):
  - Carhaix Plouguer, Carhaix-Plouguer
  - Chateauneuf du Faou, Châteauneuf-du-Faou
  - Coray, Coray
  - Guémené-sur-Scorff, Guémené-sur-Scorff
  - Guiscriff, Guiscriff
  - La Chapelle Thouarault, La Chapelle-Thouarault
  - Landeleau, Landeleau
  - Laniscat, Laniscat
  - LAZ, Laz
  - Le Faouet, Le Faouët
  - Nevez, Névez
  - Plonevez du faou, Plonévez-du-Faou
  - Plonévez du Faou, Plonévez-du-Faou
  - Plounevez-Quintin, Plounévez-Quintin
  - Plouray, Plouray
  - Poullaouen, Poullaouen
  - Rostrenen, Rostrenen
  - Roudouallec, Roudouallec
  - Saint Nicolas du Pelem, Saint-Nicolas-du-Pélem
  - Spezet, Spézet
  - Tregourez, Trégourez

IPD SHARING:
Plan to Share IPD: No